CLINICAL TRIAL: NCT01500369
Title: Effect of Remote Ischemic Preconditioning on Incidence of Atrial Fibrillation in Patients Undergoing Coronary Artery Bypass Graft Surgery A Randomized Controlled Trial
Brief Title: Effect of Remote Ischemic Preconditioning on Incidence of Atrial Fibrillation in Patients Undergoing Coronary Artery Bypass Graft Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Amir Lotfi, MD, MD, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Unique Protocol ID
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; remote ischemic conditioning
MeSH Terms: conditions — Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- remote ischemic conditiong (Active Comparator): Patients in the treatment group will receive three sequential sphygmomanometer cuff inflations on their right upper arm after induction of anesthesia in the operating room. The cuff will be inflated by the OR nurse up to 200 mmHg for five minutes each occasion, with five minutes deflation in between inflations. Following this "pre-conditioning" phase, routine anesthesia procedures will be implemented. The entire pre-conditioning phase will last 30 minutes.
  Interventions: Other: sphygmomanometer cuff inflations
- Standard Care (Placebo Comparator): Patients in the control group will have the sphygmomanometer cuff placed on their right upper arm, but the cuff will not be inflated. Similar to patients in the treatment group, patients in the control group will undergo the same 30 minute delay before induction of anesthesia and surgery
  Interventions: Other: standard of care

INTERVENTIONS:
Other: sphygmomanometer cuff inflations — : Patients in the treatment group will receive three sequential sphygmomanometer cuff inflations on their right upper arm after induction of anesthesia in the operating room. The cuff will be inflated by the OR nurse up to 200 mmHg for five minutes each occasion, with five minutes deflation in between inflations. Following this "pre-conditioning" phase, routine anesthesia procedures will be implemented. The entire pre-conditioning phase will last 30 minutes.
  Arms: remote ischemic conditiong
Other: standard of care — Placebo Comparator
  Arms: Standard Care

SUMMARY:
Atrial fibrillation is the most common arrhythmic complication after coronary artery bypass grafting (CABG). Post operative atrial fibrillation (POAF) increases morbidity and mortality. Inflammation could be a factor in POAF and recent evidence of remotely inducing ischemia may reduce inflammation and cardiac injury. The investigators plan to use a blood pressure cuff on the arm as a method to produce remote ischemia and assess the occurrence of POAF for seven day.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common arrhythmic complication after coronary artery bypass grafting (CABG) (1). It remains challenging to prevent, treat, or cure (2). It contributes to increased mortality (3), heart failure (4), stroke (5), increase in length of hospital stay, intensive care unit readmission, and treatment costs (6). The pathogenesis of atrial fibrillation (AF) after cardiac surgery is considered to be multifactorial. Some of the factors include patient's preoperative status, age, and preexisting electrocardiogram abnormalities (7). Intra-operative stress also plays key role due to occurrence of reperfusion, inflammation, oxidative stress, or hemostasis (8, 9). Post operatively, almost all AF episodes occur within the first 6 days following cardiac surgery, with the peak incidence on the second or third post-operative day which coincides with the peak of systemic inflammation caused by surgery and with atrial stretch (10).

Despite improvement in medical therapy, surgical technique, and anesthesia AF occurs in 25-40% of patients undergoing CABG (1, 11). However a recent meta-analysis demonstrated that pharmacological therapy that reduces post-operative AF, reduces length of stay, the cost of the hospitalization, and potential stroke (12). Therefore, there has been great interest to establish strategies to prevent this arrhythmia. Ischemic preconditioning is among the strategies which have shown myocardial protective effect during CABG (13). It was first described in 1986 in dog to provide a protective effect on the myocardium that is later subjected to a sustained bout of ischemia (14). Subsequently, in various clinical setting it demonstrated that ischemic preconditioning reduces the incidence of cardiac arrhythmias (15). In addition the efficacy of preconditioning in cardiac surgery and percutaneous coronary interventions has been demonstrated in human being (16).

The exact cellular mechanism of preconditioning is still controversial. Among mediators such as NO˙, ˙OH, and ONOO- which may play role in both ischemia/reperfusion injury and in the development of the cardio-protective effects of preconditioning (17); NO˙ has been considered to attenuate oxidative stress mediated cell injury during ischemia/ reperfusion. However, whether NO˙ plays a protective or detrimental role in myocardial ischemia/reperfusion injury or preconditioning remains controversial (18, 19). In a recent study, Jannati et al. demonstrated that myocardial ischemic preconditioning by aortic cross clamping in patients undergoing CABG reduced the incidence of post operative AF (20).

Currently there is no clinical preconditioning protocol or tool being utilized during CABG. Additionally, aortic cross clamping may increase the risk of embolic stroke, particularly in elderly patients (21). Therefore, we are conducting a prospective single-blinded randomized controlled study to demonstrate whether remote ischemic preconditioning reduces incidence of post operative AF.

IV. RESEARCH DESIGN

OBJECTIVE: To investigate if remote ischemic preconditioning will reduce the risk of post operative atrial fibrillation in patient undergoing elective CABG.

Study Population

This will be a prospective randomized controlled study on patients older than 18 years old who are undergoing elective CABG with or without valve surgery at Baystate Medical Center. Exclusion criteria include any preoperative rhythm other than sinus, history of atrial fibrillation, New York Hear Association (NYHA) IV congestive heart failure, cardiogenic shock, emergent CABG and/or valve surgery, bleeding diathesis, and women of child-bearing potential. Eligible patients will participate after obtaining consent. Patients will be blindly randomize patient into two groups:

Study Groups

1. Treatment Group: Patients in the treatment group will receive three sequential sphygmomanometer cuff inflations on their right upper arm after induction of anesthesia in the operating room. The cuff will be inflated by the OR nurse up to 200 mmHg for five minutes each occasion, with five minutes deflation in between inflations. Following this "pre-conditioning" phase, routine anesthesia procedures will be implemented. The entire pre-conditioning phase will last 30 minutes.
2. Control Group: Patients in the control group will have the sphygmomanometer cuff placed on their right upper arm, but the cuff will not be inflated. Similar to patients in the treatment group, patients in the control group will undergo the same 30 minute delay before induction of anesthesia and surgery.

Data Collection After completion of surgery, the telemetry monitor for atrial fibrillation will be reviewed daily and 12-lead electrocardiography will be obtained as needed. All episodes of atrial fibrillation on telemetry will be collected, reviewed, and entered in a data sheet. The data sheet will be available in the chart of all patients enrolled in the study (study and control groups). These data will be transferred and will be kept in a data set which will be coded with a study ID number. The identifiers will include age, sex, medical record number (MRN), date of admission, date of discharge, and length of post operative hospital stay. We will collect baseline characteristic including age, diabetes mellitus, hypertension, myocardial infarction, left ventricular ejection fraction, concomitant valvular disease, history of heart surgery, medications, type of surgery, and post-operation atrial fibrillation. Data collection will be closed at the end of one-year and will be presented for publication or presentation, while no patient will be identified.

Subject Confidentiality To maintain patient confidentiality, all the collected data will be in a password protected computer and all the paper files will be kept in a locked cabinet in the PIs office. All data will be entered in a spreadsheet and will be immediately de-identified by creating a study ID number. The master list containing patient ID code will be in a password protected computer.

Outcome Events The primary outcome will be atrial fibrillation lasting for five minutes or longer during the first seven days after surgery. Secondary outcomes include length of hospital stay, incidence of myocardial infraction, stroke, and postoperative day of arrhythmic event.

EKG recording Twelve-lead electrocardiograms will be recorded preoperatively, following surgery on return to the intensive care unit, and daily during their first seven days of hospital stay. Also the arrhythmic events will be recorded through telemetry during hospital stay.

Randomization Procedure Once eligibility has been established and consent has been obtained, patients will be randomized according to computer generated randomization procedure. Patients will be randomized in blocks sizes of 4 and 6. Permuted block randomization will insure that study groups will remain balanced at the completion of each block and that unbalanced study groups is minimized if the study is terminated during a block interval.

Data analysis Treatment and control groups will be compared on baseline characteristics to identify patient or clinical factors that may not have been adequately balanced by the randomization procedure. Continuous variables will be compared using 2-sample t-tests or its non-parametric equivalent (Wilcoxon rank-sum test), while categorical variables will be compared using Pearson chi-square or Fisher's exact test. Differences on baseline characteristics achieving a p-value of .15 or less will be included in subsequent multivariable analysis. Multivariable analyses will be conducted using logistic regression. The dependent variable will be the dichotomous variable of the presence or absence of atrial fibrillation at any time during the 7-day follow-up period. Independent variables will include the dichotomous variable representing study group, as well as baseline characteristics requiring adjustment. Data will be analyzed on an intention-to-treat basis.

Sample Size The sample size was calculated on an estimated 35% incidence atrial fibrillation over the 7-day period in control patients undergoing CABG. To detect an absolute reduction of 13 percentage points (i.e., 35% in the control group vs. 22% in the treatment group) at 5% significance and 80% power, the study requires randomization of 205 patients per study group.

Early Termination of Study To determine whether early termination of the trial is necessary due to larger than expect benefit or larger than expected harm, we plan one interim look at the data when 50% of the patients have completed follow-up. We use the Obrien-Fleming (1979) spending function to adjust the alpha comparison at the interim analysis and the final analysis in order to maintain an overall critical level of 5% (overall p-value is 5%). Thus, the trial will be terminated early if the at the interim analysis the absolute difference in the proportion of atrial fibrillation between the study groups achieves a significance level of p ≤ 0.003. For the final analysis at study completion, significance testing will be conducted at p ≤ 0.047. This adjustment insures that the comparisons will be conducted at an overall significance level of 5%.

Budget No expenses are anticipated.

Disclosures Patient confidentiality will be ensured by coding all the data. No direct patient contact. No active intervention affecting patient care or health is proposed. No vulnerable groups are included in the study. Patient consent would not be required for inclusion in the study. None of the investigators have a vested interest in the outcome/s of this study that may affect their objectivity in data gathering/analysis or the recommendations they make based on the results of the study.

Risk benefit ratio Minimal risk is involved with this study. However, by demonstrating the benefit of non-invasive remote ischemic preconditioning in reducing the incident of post operative atrial fibrillation we will add new information to the literature. More importantly, another preventive option will be available in reducing the incidence of post operative atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* This will be a prospective randomized controlled study on patients older than 18 years old who are undergoing elective CABG with or without valve surgery.

Exclusion Criteria:

* any preoperative rhythm other than sinus,
* history of atrial fibrillation,
* New York Hear Association (NYHA) IV congestive heart failure,
* cardiogenic shock,
* emergent CABG and/or valve surgery,
* bleeding diathesis, and
* women of child-bearing potential. Eligible patients will participate after obtaining consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Post op atrial fibrillation | 7 days post cardiac surgery
  Assess the indicence of post operative atrial fibrillation

SECONDARY OUTCOMES:
Stroke | 7 days
  Post operative stroke

CONTACTS AND LOCATIONS:
Overall Officials: amir Lotfi, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States